## The Effects of α-Tocopherol in Hemolysis and Oxidative Stress Marker

## on Red Cell Membrane β-Thalassemia Major

**Background:** The accumulation of unpaired  $\alpha$ -globin chains in  $\beta$ -thalassemia major patients may clinically create ineffective erythropoiesis, hemolysis, and chronic anemia. Multiple blood transfusions and iron overload cause cellular oxidative damage. However,  $\alpha$ -tocopherol, an antioxidant, has been known as a potent scavenger of lipid radicals in the red cell membrane of  $\beta$ -thalassemia major patients.

**Purpose:** To evaluate the effects of  $\alpha$ -tocopherol in hemolysis and oxidative stress on the red cell membrane of  $\beta$ -thalassemia major.

**Methods:** In this randomized controlled trial, we allocated subjects in the placebo and  $\alpha$ -tocopherol groups. Doses of  $\alpha$ -tocopherol were based on the recommendation of Institute of Medicine: 4–8 years old 200 mg/day; 9–13 years old 400 mg/day; 14–18 years old 600 mg/day. Hemolysis, oxidative stress, and antioxidant variables were evaluated before and after 4 weeks of consuming either  $\alpha$ -tocopherol or placebo, performed prior to blood transfusions.

Figure. Study Protocol

